CLINICAL TRIAL: NCT06029478
Title: Understanding Engagement Trends in Chondrosarcoma Clinical Trials: Investigating Participation Patterns Among Chondrosarcoma Patients
Brief Title: Understanding Engagement Trends in Chondrosarcoma Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84518615
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Chondrosarcoma
Keywords: chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical research usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of chondrosarcoma patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future chondrosarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Able to comprehend the investigational nature of the protocol and provide informed consent
* Diagnosis of chondrosarcoma

Exclusion Criteria:

* No diagnosis of chondrosarcoma confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chondrosarcoma who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of chondrosarcoma patients who decide to enroll in a clinical trial | 3 months
Rate of chondrosarcoma patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Speetjens FM, de Jong Y, Gelderblom H, Bovee JV. Molecular oncogenesis of chondrosarcoma: impact for targeted treatment. Curr Opin Oncol. 2016 Jul;28(4):314-22. doi: 10.1097/CCO.0000000000000300. PMID 27166664
- [Background] Beena D, Kattoor J, Mathews A, P Nair S, M V, T P, N G. Mesenchymal Chondrosarcoma-A Retrospective study. Gulf J Oncolog. 2021 Jan;1(35):54-58. PMID 33716213
- [Background] Thompson LD, Gannon FH. Chondrosarcoma of the larynx: a clinicopathologic study of 111 cases with a review of the literature. Am J Surg Pathol. 2002 Jul;26(7):836-51. doi: 10.1097/00000478-200207000-00002. PMID 12131151

DOCUMENTS (1):
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT06029478/ICF_000.pdf